CLINICAL TRIAL: NCT05363826
Title: Phase I Study of the Safety of Intracavitary Photodynamic Therapy (PDT) of the Brain Bordering Resected Recurrent Glioblastoma or Gliosarcoma Using Intravenous Photobac® and a Balloon Light Applicator
Brief Title: Intracavitary Photodynamic Therapy as an Adjuvant to Resection of Glioblastoma or Gliosarcoma Using IV Photobac®
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Photolitec LLC (Industry)
Collaborators: Roswell Park Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14598; 4R44CA247127-02 (NIH)
Record Dates: First submitted 2022-04-13; First posted 2022-05-06 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma Multiforme of Brain; Glioma, Sarcomatous
Keywords: Photochemo Therapy; Photo Dynamic Therapy; PDT
MeSH Terms: conditions — Gliosarcoma

STUDY DESIGN:
Intervention Model Description: This is a phase I Drug study of the photochemotherapy drug Methyl bacteriopurpurinimide Bacteriopurpurinimide-methyl ester (registered trade name Photobac®) in adult subjects with recurrent diagnosed glioblastoma or gliosarcoma.
  We are evaluating the safety of this photosensitizing drug in an 8 step dose escalation with 3 patients per step and a fixed light dose (50 joules / square centimeter) by way of intraoperative cavitary photodynamic therapy using a balloon and spherical diffuser to deliver the light.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Photochemotherapy as an adjuvant to surgical resection of glioblastoma (Experimental): 3-(1-Butyloxy)ethyl-3-deacetyl-bacteriopurpurin-18-n-butylimide methyl ester (Photobac®) is injected 24 hours prior to surgical resection of a recurrent Glioblastoma or gliosarcoma. Immediately following the resection the cavity is treated with 50 joules/ square cm of 787 nm light .The drug dose is escalated using three patient cohorts until a dose limiting toxicity is reached or the upper limit of the 8 step escalation is reached.
  Interventions: Combination Product: photochemotherapy using 3-(1-Butyloxy)ethyl-3-deacetyl-bacteriopurpurin-18-n-butylimide methyl ester(Photobac®)

INTERVENTIONS:
Combination Product: photochemotherapy using 3-(1-Butyloxy)ethyl-3-deacetyl-bacteriopurpurin-18-n-butylimide methyl ester(Photobac®) — Intravenous injection of Photobac® 24 hours before surgical removal of recurrent GBMF.
  Immediately after resection, the cavity will be treated with 50 joules/ square cm of 787nm light. This treatment will add a maximum of 50 minutes to the surgery
  Other Names: Photobac® PDT

SUMMARY:
This study is the first step in testing the hypothesis that adding Photobac® Photodynamic Therapy to surgical removal of a glioblastoma or gliosarcoma will be both safe and effective.

Photodynamic Therapy (PDT) combines light and a photosensitizer. PDT has been used to treat a variety of cancers with varying degrees of success.

For the past thirty years Photolitec has been working to develop a treatment for glioblastoma or gliosarcoma using light and a photosensitizer. Photolitec's scientists were looking for a photosensitizer that:

1. has no significant systemic toxicity apart from some temporary skin photosensitivity,
2. crosses the blood brain barrier,
3. accumulates to a high level in glioblastoma and minimally in the brain,
4. is activated by the wavelength of light that penetrates most deeply into the brain,
5. minimizes any temporary skin photosensitivity.

Preliminary testing indicates the Photolitec team has achieved these five goals. Photolitec is now able to offer a clinical trial based on the results of this work.

DETAILED DESCRIPTION:
Twenty four hours before surgery the patient will receive an intravenous injection of Photobac®. This will make the brain tumor sensitive to light. Lighting up the brain using a low power near infrared laser will kill cells that contain Photobac®.

Photobac® crosses the blood brain barrier. Compared to the brain at 24 hours after injection, the tumor holds significantly more Photobac®. This Selective retention by tumors is the reason PDT has proved a valuable weapon against other types of tumors.

Once the surgeon has removed the tumor as completely as possible, the brain that bordered the tumor will be illuminated with near infrared light from a low power laser. This will destroy tumor cells hiding deep in the brain. Such cells cause tumor recurrence.

The light treatment will add about one hour to the surgery. The Patient will be asleep during this procedure. The patient will receive standard post-surgical care during recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18years.
2. Subject has a Karnofsky performance status ≥ 70 (i.e. the subject must be able to care for himself/herself with occasional help from others; refer to Appendix G).
3. Subject has pathologically confirmed diagnosis of glioblastoma or gliosarcoma.
4. Subject has recurrent or progressive tumor following standard therapy.
5. Subject has recurrent cerebral tumor that in the opinion of the treating neurosurgeon is surgically resectable.
6. Subject has the following clinical laboratory values obtained within 14 days prior to registration:

   Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L Hemoglobin (Hgb) > 9.0 g/dL Plasma total bilirubin: ≤ 1.5 x ULN ALT and AST ≤ 2.0 x ULN Creatinine clearance >60 WBC ≥ 4000 INR ≤ 1.1 x ULN
7. Subject will have been off all anticoagulant therapy (e.g., warfarin, heparin, enoxaparin, rivaroxaban, apixaban, aspirin) for at least 5 days before surgery and Photobac® infusion.
8. No active bleeding or pathological condition that in the judgement of the principal investigator carries a high risk of bleeding
9. Subject of child-bearing potential "agrees to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and have a negative pregnancy test prior to starting study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
10. Subject has completed radiation therapy (RT) and temozolomide (TMZ) for the treatment of their glioblastoma or gliosarcoma at least 30 days prior to entry
11. Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

1. Subject has serious concurrent infection or medical illness, which in the treating physician's opinion would jeopardize the ability of the subject to receive the treatment outlined in this protocol with reasonable safety.
2. Subject is pregnant or breast-feeding.
3. Subject has latex allergy.
4. Subject has received another chemotherapeutic or investigational agent in addition to radiation therapy and concomitant temozolomide treatment within 30 days of planned PDT.
5. Subject has persistent toxicity of prior therapy.
6. Subject has gliomatosis cerebri.
7. Subject has cerebral tumor that in the opinion of the treating neurosurgeon is unresectable.
8. Subject has brainstem, spinal cord or cerebellar involvement by tumor.
9. Subject has known human immunodeficiency virus (HIV) positivity or acquired immunodeficiency syndrome (AIDS) related illness or other serious medical illness.
10. Subject has contraindication to MRI scans or gadolinium contrast agent.
11. Subject has history of porphyria, hypersensitivity to porphyrin or porphyrin-like compounds or any other abnormal skin photosensitivity.
12. Subject is unwilling or unable to follow protocol requirements.
13. Subject has any condition which in the Investigator's opinion makes the subject unsuitable to receive the study drug. Must be reported.
14. Subject has any condition which in the treating neurosurgeon's opinion makes the subject unsuitable to undergo craniotomy for tumor resection.
15. Subject has received an investigational agent within 30 days prior to planned PDT.
16. Subject has midline shift > 1 cm.
17. Subject is unable to give consent to participate in the study.
18. Subject has a QTC interval > 470 milliseconds (CTCAE grade 1) using Frederica's QT correction formula.
19. Subject has serious concurrent infection or medical illness, which in the treating physician's opinion would jeopardize the ability of the subject to tolerate the added hour o anesthesia outlined in this protocol with reasonable safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity will be measured using CTCAE v5 ( Common Terminology Criteria for Adverse Events | .up to 24 hours
  •A dose limiting toxicity (DLT)will stop the escalation. A DLT includes all greater than or equal to grade 3 non-hematological toxicities and all greater than or equal to grade 4 hematological toxicities per CTCAE v 5.0
The Maximum Tolerable drug Dose (MTD) will be determined by evaluating the safety of a fixed light dose and escalating drug dose | up to one week
  The MTD will be determined by first discovering the dose limiting toxicity ( DLT). As defined above and following the procedure for determining the MTD from the DLT found in the protocol. It is expected that the DLT may be acute neurotoxicity caused by brain swelling.
Measure the Photobac concentration in blood. | up to12 weeks
  Photobac® concentration in blood will be measured by drawing blood at various time points. The blood will be spun down and the concentration in the serum measured spectroscopically. Non-linear regression will be used to determine the clearance rate constants from these data.
Measure Photobac® concentration in tumor tissue removed during resection and in the bed of the tumor both before and after ligh treatment. | 1 hour
  The tissue samples will be subject to chemical extraction of the Photobac®. Photobac® concentration in the extract will be measured spectroscopically.
Time of Progression Free Survival | up t o18 months
  The duration of progression free survival will be assessed by a Roswell neuroradiologist using RANO criteria.
Overall survival from time of diagnosis | up to 18 months
  Patients will be followed for the duration of the study and if possible until death.

SECONDARY OUTCOMES:
Duration and severity of skin photosensitivity t osimulated sunlight . | 1 week
  If the patient's condition permits, a solar simulator will be used to assess the patient's skin photosensitivity .The severity and duration of sensitivity will be assessed using the Draize scale. The Draize scale ranges from zero indicating no reaction to 4 indicating a severe reaction. Two numbers will be reported one for erythema and the second for edema
Assess patterns of treatment failure for any association with the drug dose | up to 15 months.
  Duration of survival and progression free survival will be examined for evidence of a Photobac® dose dependant response.
Measure Stat 3 Crosslinking as a quantitative marker of singlet oxygen tissue damage | 1 hour
  The samples of tissue taken from the tumor bed will be assayed for the degree of stat 3 crosslinking. Stat3 crosslinking is caused by singlet oxygen damage and is expected correlate with the PDT dose.

CONTACTS AND LOCATIONS:
Overall Officials: William R Potter, MA, Principal Investigator — Photolitec LLC; Robert Fenstermaker, MD, Principal Investigator — Roswell Park Dept of Neurosurgery
Locations (1):
- Roswell Park Cancer, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel N, Pera P, Joshi P, Dukh M, Tabaczynski WA, Siters KE, Kryman M, Cheruku RR, Durrani F, Missert JR, Watson R, Ohulchanskyy TY, Tracy EC, Baumann H, Pandey RK. Highly Effective Dual-Function Near-Infrared (NIR) Photosensitizer for Fluorescence Imaging and Photodynamic Therapy (PDT) of Cancer. J Med Chem. 2016 Nov 10;59(21):9774-9787. doi: 10.1021/acs.jmedchem.6b00890. Epub 2016 Oct 31. PMID 27749069